CLINICAL TRIAL: NCT04342897
Title: A Randomized, Double-blind, Placebo-controlled, Clinical Trial of LY3127804 in Patients Who Are Hospitalized With Pneumonia and Presumed or Confirmed COVID-19
Brief Title: A Study of LY3127804 in Participants With COVID-19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial terminated for futility.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17824; I7W-MC-UDAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-04-10; First posted 2020-04-13 (Actual); Results first posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: COVID-19; Pneumonia
Keywords: Corona Virus Disease 19 (COVID-19); 2019 Novel Coronavirus (2019 n-COV); Severe Acute Respiratory Syndrome (SARS); Pulmonary Disease; SARS-CoV-2
MeSH Terms: conditions — COVID-19; Pneumonia; Severe Acute Respiratory Syndrome; Lung Diseases | interventions — zansecimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3127804 (Experimental): Participants received 20 milligrams (mg) per kilogram (kg) of LY3127804 as an intravenous (IV) infusion on Days 1 and 15.
  Interventions: Drug: LY3127804
- Placebo (Placebo Comparator): Participants received 20 mg/kg of Placebo as an IV infusion on Days 1 and 15.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3127804 — Administered IV
  Arms: LY3127804
Drug: Placebo — Administered IV
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled, clinical trial of LY3127804 in participants who are hospitalized with pneumonia and presumed or confirmed COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Are hospitalized with pneumonia, and presumed or confirmed COVID-19
* Are able and willing to give signed informed consent (legally authorized representative can provide informed consent if needed)

Exclusion Criteria:

* Female participants must not be pregnant and/or lactating
* Have Acute Respiratory Distress Syndrome (ARDS) or will require immediate intermittent mandatory ventilation (IMV), or are ineligible for IMV
* Have any concurrent serious medical condition (for example dialysis) or concomitant medication that would preclude participation in the study
* Are moribund irrespective of the provision of treatments
* Have a known history or show evidence of human immunodeficiency virus (HIV) and/or hepatitis
* Have recently undergone major surgery or central venous access device placement
* Have a significant bleeding disorder or active vasculitis
* Have experienced a thromboembolic event
* Have symptomatic congestive heart failure, or symptomatic or poorly controlled cardiac arrhythmia
* Have a serious, nonhealing wound, peptic ulcer, or bone fracture
* Have liver cirrhosis
* Have a known sensitivity to monoclonal antibodies (mAbs) or other therapeutic proteins
* Have a history of hypertensive crisis or hypertensive encephalopathy or current, poorly controlled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-10-12 (Actual); Study Completion 2020-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (13):
- United States (13):
  - Banner Univ Med Ctr Phoenix, Phoenix, Arizona
  - Banner Univ Med Ctr Tucson, Tucson, Arizona
  - National Jewish Medical and Research Center, Denver, Colorado
  - Nuvance Danbury Hospital, Danbury, Connecticut
  - NorthShore University HealthSystem, Evanston, Illinois
  - Parkview Research Center, Fort Wayne, Indiana
  - Franciscan St. Francis Health, Indianapolis, Indiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Henry Ford Hospital Detroit, Detroit, Michigan
  - Allina Hospital Network, Minneapolis, Minnesota
  - State University of New York Hospital, Syracuse, New York
  - East Carolina University, Greenville, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting
Access Criteria: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting
URL: http://vivli.org/

REFERENCES:
- [Derived] Jones RS, Smith PS, Berg PH, de la Pena A, Cook PP, Shawa I, Kioussopoulos KM, Hu Y, Schott RJ. Efficacy and Safety of LY3127804, an Anti-Angiopoietin-2 Antibody, in a Randomized, Double-Blind, Placebo-Controlled Clinical Trial in Patients Hospitalized with Pneumonia and Presumed or Confirmed COVID-19. Clin Med Insights Circ Respir Pulm Med. 2022 Aug 10;16:11795484221119316. doi: 10.1177/11795484221119316. eCollection 2022. PMID 35991210
- See also: A Study of LY3127804 in Participants With COVID-19 — https://www.lillytrialguide.com/en-US/studies/covid-19--coronavirus-/UDAA#?postal=

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LY3127804 | Placebo
Started | 47 | 48
Received at Least One Dose of Study Drug | 47 | 48
Completed | 33 | 36
Not Completed | 14 | 12
Not completed — Death | 7 | 4
Not completed — Lost to Follow-up | 6 | 6
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug.
Groups:
- LY3127804: Participants received 20 mg/kg of LY3127804 as an IV infusion on Days 1 and 15.
- Total: Total of all reporting groups
Arm/Group | LY3127804 | Placebo | Total
Number analyzed (Participants) | 47 | 48 | 95
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.3 (14.13) | 55.5 (14.40) | 54.9 (14.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 29 | 31 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 20 | 43
  Not Hispanic or Latino | 24 | 28 | 52
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 8 | 7 | 15
  White | 36 | 38 | 74
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 47 | 48 | 95
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 33.74 (6.963) | 33.70 (7.715) | 33.72 (7.314)

OUTCOME MEASURES:

1. Primary Outcome: Ventilator Free Days
Description: Ventilator-free days were defined as the number of days from Day 1 through Day 28 on which a participant breathed without assistance, if the period of unassisted breathing lasted at least 24 consecutive hours and the participant did not die within 28 days from the first dose of the study drug.
Time Frame: Day 1 through Day 28
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: days
Arm/Group | LY3127804 | Placebo
Number analyzed (Participants) | 47 | 48
days | 28 [12 to 28] | 28 [4 to 28]

2. Secondary Outcome: Number of Participants Reported Lowest Score on National Institute of Allergy and Infectious Diseases (NIAID) Ordinal Scale
Description: The NIAID ordinal scale clinical status was defined as the lowest score achieved for that day, the lowest NIAID score from Day 1 through Day 28 for each participant was reported. NIAID ordinal assessment levels are reported by using the following 8 point scale, where a higher score is a better outcome: 1) death, 2) hospitalized, on invasive mechanical ventilation (IMV) or extracorporeal membrane oxygenation (ECMO), 3) hospitalized, on non-invasive ventilation or high-flow oxygen devices, 4) hospitalized, requiring supplemental oxygen, 5) hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19-related or otherwise), 6) hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care, 7) not hospitalized, limitation on activities and/or requiring home oxygen, and, 8) not hospitalized, no limitations on activities.
Time Frame: Day 1 through Day 28
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | LY3127804 | Placebo
Number analyzed (Participants) | 47 | 48
Participants
  NIAID Level 1 | 7 | 4
  NIAID Level 2 | 3 | 2
  NIAID Level 3 | 12 | 21
  NIAID Level 4 | 24 | 19
  NIAID Level 5 | 1 | 2
  NIAID Level 6 | 0 | 0
  NIAID Level 7 | 0 | 0
  NIAID Level 8 | 0 | 0

3. Secondary Outcome: Percentage of Participants With Complete Response
Description: Complete response was defined as being alive and never requiring mechanical ventilator support (at any point while on study) through Day 28.
Time Frame: Day 1 through Day 28
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | LY3127804 | Placebo
Number analyzed (Participants) | 47 | 48
percentage of participants | 78.7 | 87.5

4. Secondary Outcome: Number of Participants Who Died Between Day 1 Through Day 28
Time Frame: Day 1 through Day 28
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | LY3127804 | Placebo
Number analyzed (Participants) | 47 | 48
participants | 7 | 4

5. Secondary Outcome: Length of Hospitalization
Description: Days of participants hospitalization.
Time Frame: Day 1 through Day 28
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | LY3127804 | Placebo
Number analyzed (Participants) | 47 | 48
days | 6 [4 to 12] | 6 [5 to 13.5]

6. Secondary Outcome: Number of Participants With Treatment-Emergent Serious Adverse Events (TE-SAE)
Description: An SAE is any AE from this study that results in one of the following outcomes: death that is not related to COVID-19 or a sequela of COVID-19 or death that is considered by the investigator to be related to study drug, prolonged inpatient hospitalization or re-hospitalization life-threatening experience (that is, immediate risk of dying), persistent or significant disability/incapacity, congenital anomaly/birth defect, important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require intervention to prevent one of the other SAE outcomes.
Time Frame: Day 1 through Day 60
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | LY3127804 | Placebo
Number analyzed (Participants) | 47 | 48
participants | 6 | 2

7. Secondary Outcome: Number of Participants With Any Treatment Emergent Adverse Event (TEAE)
Description: TEAE was defined as any untoward medical occurrence that emerges during a defined treatment period, having been absent pre-treatment, or worsens relative to the pretreatment state, and does not necessarily had a causal relationship with the study treatment.
Time Frame: Day 1 through Day 60
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | LY3127804 | Placebo
Number analyzed (Participants) | 47 | 48
participants | 33 | 31

ADVERSE EVENTS:
Time Frame: Day 1 through Day 60
Description: All randomized participants who received at least 1 dose of study drug.
Arm/Group | LY3127804 | Placebo
All-Cause Mortality (participants affected / at risk) | 8/47 | 6/48
Serious Adverse Events (participants affected / at risk) | 6/47 | 2/48
Other Adverse Events (participants affected / at risk) | 30/47 | 31/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY3127804 (N=47) | Placebo (N=48)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY3127804 (N=47) | Placebo (N=48)
Leukocytosis (Blood and lymphatic system disorders) | 5 (5) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (6) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Oral candidiasis (Infections and infestations) | 3 (3) | 0 (0)
Septic shock (Infections and infestations) | 3 (3) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (6) | 3 (3)
Encephalopathy (Nervous system disorders) | 3 (3) | 2 (3)
Anxiety (Psychiatric disorders) | 4 (4) | 6 (6)
Insomnia (Psychiatric disorders) | 5 (5) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 4 (6)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Hypertension (Vascular disorders) | 4 (5) | 3 (3)
Hypotension (Vascular disorders) | 3 (4) | 3 (4)

LIMITATIONS AND CAVEATS:
The study was terminated for futility reason.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/97/NCT04342897/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/97/NCT04342897/SAP_001.pdf